CLINICAL TRIAL: NCT07260474
Title: Comparison of the Amplatzer Amulet Versus LAmbre Device for Left Atrial Appendage Closure: the CALAMBRE Randomized Clinical Trial
Brief Title: Comparison of the Amplatzer Amulet Versus LAmbre Device for Left Atrial Appendage Closure
Acronym: CALAMBRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC48-CALAMBRE
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amplatzer Amulet™left atrial appendage occluder (Other)
  Interventions: Device: Patients implanted with Amplatzer Amulet™
- LAmbre™left atrial appendage occluder (Other)
  Interventions: Device: Patients implanted with LAmbre™

INTERVENTIONS:
Device: Patients implanted with Amplatzer Amulet™ — Left atrial appendage closure with the Amplatzer Amulet™ device. The procedure will be performed according to standard practice using the manufacturer's instructions for use.
  Arms: Amplatzer Amulet™left atrial appendage occluder
Device: Patients implanted with LAmbre™ — Left atrial appendage closure with the LAmbre™ device. The procedure will be performed according to standard practice using the manufacturer's instructions for use.
  Arms: LAmbre™left atrial appendage occluder

SUMMARY:
Clinical investigation with CE-marked medical devices, multicenter, prospective, randomized and controlled. Patients with non-valvular atrial fibrillation at high embolic risk and with at least one high bleeding risk criterion according to the Munich consensus document will be randomized to left atrial appendage closure with either the Amplatzer Amulet™ or the LAmbre™ device. The study is designed to compare the efficacy and safety of both devices regarding successful implantation, effective appendage closure, and clinical outcomes at follow-up.

DETAILED DESCRIPTION:
Clinical investigation with CE-marked medical devices, multicenter, prospective, randomized and controlled. Patients with non-valvular atrial fibrillation at high embolic risk and with at least one high bleeding risk criterion according to the Munich consensus document will be randomized to left atrial appendage closure with either the Amplatzer Amulet™ or the LAmbre™ device. The study is designed to compare the efficacy and safety of both devices regarding successful implantation, effective appendage closure, and clinical outcomes at follow-up.

ELIGIBILITY:
Inclusion Criteria:

(MUST MEET ALL INCLUSION CRITERIA)

* Patient with aged ≥18 years AND;
* Patient have non-valvular atrial (NVAF) with a CHA2DS2-VASc score ≥2, and presented at least one high-bleeding-risk criterion according to the Munich consensus document AND;
* Patient are required to undergo preprocedural TEE / CCTA to confirm the absence of LAA thrombus and to ensure that LAA anatomy is suitable for closure with either device.
* Patient who has been informed of the characteristics of the study and has provided written informed consent..

Exclusion Criteria:

(MUST NOT MEET ANY EXCLUSION CRITERIA)

* Patient life expectancy <1 year (terminal illness).
* Patient with requirement for oral anticoagulation therapy for any indication other than non-valvular atrial fibrillation.
* Patient with prior surgical ligation or obliteration of the left atrial appendage.
* Patient with history of allergic reaction or intolerance to any material used in the study devices or to any of the antithrombotic agents required post-procedure.
* Patient with active systemic infection.
* Patient with concurrent participation in another investigational study that may affect study results.
* Patient with inability or unwillingness to comply with the study protocol or follow-up requirements.
* Patient pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: Device success | 3 months
  Percentage Device success defined as: Successful deployment and stable implantation of the assigned device within the left atrial appendage during the index procedure and no crossover to the alternative device and effective closure of the appendage with a residual leak ≤5 mm as assessed by TEE(Transesophageal Echocardiography) or CCTA (Cardiac Computed Tomography Angiography) at 90 days.

SECONDARY OUTCOMES:
SAFETY: Clinical success | 3 months
  Percentage of Device success plus absence of all-cause mortality, stroke, systemic embolism, or procedure-related complications at 90 days.
SAFETY: Procedure-related complications | 7 days
  Percentage of Composite of death, stroke, systemic or pulmonary embolism, air embolism, any bleeding, pericardial effusion, vascular access complication, device-related complication, or AKI (Acute Kidney Injury) within 7 days (or later if related to the procedure).
EFFICACY: Residual leak | 3 months
  Percentage of residual leak >5 mm as assessed by TEE or CCTA (core lab evaluation).
EFFICACY: Residual leak | 12 months
  Percentage of residual leak >5 mm as assessed by TEE or CCTA (core lab evaluation).
SAFETY:Device-related thrombus (DRT) | 3 months
  Percentage of Homogeneous mass (TEE) or hypoattenuated thickening (CCTA) on the atrial surface of the device, adjudicated by independent imaging experts.
SAFETY: MACE | 3 months
  Percentage of Composite of all-cause mortality, cardiovascular mortality, ischemic or hemorrhagic stroke, systemic embolism, pulmonary embolism, myocardial infarction, and bleeding (classified by BARC (Bleeding Academic Research Consortium)).
SAFETY: MACE | 12 months
  Percentage of Composite of all-cause mortality, cardiovascular mortality, ischemic or hemorrhagic stroke, systemic embolism, pulmonary embolism, myocardial infarction, and bleeding (classified by BARC (Bleeding Academic Research Consortium)).

REFERENCES:
- [Background] Landmesser U, Skurk C, Tzikas A, Falk V, Reddy VY, Windecker S. Left atrial appendage closure for stroke prevention in atrial fibrillation: current status and perspectives. Eur Heart J. 2024 Aug 21;45(32):2914-2932. doi: 10.1093/eurheartj/ehae398. PMID 39027946
- [Background] Lakkireddy D, Ellis CR, Thaler D, Swarup V, Gambhir A, Hermiller J, Nielsen-Kudsk JE, Worthley S, Nair D, Schmidt B, Horton R, Gupta N, Anderson JA, Zhao H, Alkhouli M, Windecker S. 5-Year Results From the AMPLATZER Amulet Left Atrial Appendage Occluder Randomized Controlled Trial. J Am Coll Cardiol. 2025 Mar 25;85(11):1141-1153. doi: 10.1016/j.jacc.2024.10.101. Epub 2024 Nov 18. PMID 39570242
- [Background] Alkhouli M, Freeman JV, Ellis CR, Shah AP, Gada H, Coylewright M, Lo M, Makkar A, Agarwal H, Lakkireddy D. First Experience With Amulet in the United States: Early Insights From EMERGE LAA Postapproval Study. JACC Cardiovasc Interv. 2024 Jan 19:S1936-8798(23)01553-4. doi: 10.1016/j.jcin.2023.11.027. Online ahead of print. PMID 38310499
- [Background] Bangash AB, Li Y, Huang W, Zhong J, Zheng H, Zhang D, Zeng A, Wang R, Zhao W, Wang M, Zhao Y, Yu L, Liu Q, Jiang R, Jiang C, Zhang J. Left atrial appendage occlusion using the LAmbre device in atrial fibrillation patients with a history of ischemic stroke: 1-Year outcomes from a multicenter study in China. Pacing Clin Electrophysiol. 2023 Dec;46(12):1478-1483. doi: 10.1111/pace.14866. Epub 2023 Nov 9. PMID 37943004
- [Background] Samaras A, Papazoglou AS, Balomenakis C, Bekiaridou A, Moysidis DV, Patsiou V, Orfanidis A, Giannakoulas G, Kassimis G, Fragakis N, Saw J, Landmesser U, Alkhouli MA, Tzikas A. Residual leaks following percutaneous left atrial appendage occlusion and outcomes: a meta-analysis. Eur Heart J. 2024 Jan 14;45(3):214-229. doi: 10.1093/eurheartj/ehad828. PMID 38088437